CLINICAL TRIAL: NCT03583411
Title: Platelets Count Alterations in Patients With Acute Coronary Syndrome: Epidemiology and Prognostic Role
Brief Title: Platelets Count Alterations in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S_23_10_17_2001
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Acute Coronary Syndrome
Keywords: thrombocytopenia; thrombocytosis
MeSH Terms: conditions — Acute Coronary Syndrome; Thrombocytopenia; Thrombocytosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute coronary syndrome (ACS) patients: ACS subjects hospitalized in the Cardiology 1 - UTIC department of ASST Grande Ospedale Metropolitano Niguarda between 2014 and 2017
  Interventions: Other: Epidemiological data collection

INTERVENTIONS:
Other: Epidemiological data collection — To profile each subject enrolled in the study, anamnesis and different personal, clinical, procedural, pharmacological and follow up related variables will be collected. Data collection, maintenance and analysis will be performed using a database that will be developed, managed and updated by study promoter, in accordance with Good Clinical Practice (GCP)

SUMMARY:
Platelet count alterations (thrombocytopenia and thrombocytosis) are a common condition in patients hospitalised for acute coronary syndrome (ACS), both at disease onset and in the following recovery phase.1-3 Different factors can explain this phenomenon. Thrombocytopenia could be either due to neurohormonal activation and the inflammatory process following myocardial necrosis leading to increased macrophage activation with increased clearance of platelets, or to an immuno-modulated mechanism caused by the administration of antiaggregant/anticoagulant drugs (heparin, glycoprotein IIb/IIIa inhibitors, P2Y12 inhibitors).

Even the invasive treatment of coronaropathy during hospitalization, with angioplasty and stent implantation procedures and/or the eventual implantation of temporary mechanical blood circulation assistant devices [aortic counterpulsation, Impella, ECMO (Extracorporeal Membrane Oxygenation)], could further favour the phenomenon.4 Vice versa, thrombocytosis occurring during ACS has a reactive origin, caused by increased IL-6 production which, in turn, leads to an increase in thrombopoietin formation in the liver, causing a consequent stimulatory activity on megakaryocytes.2 Different studies have demonstrated a significant correlation between platelets count disorders and patient outcome (survival during hospitalization and in the immediate follow-up).5-11 This association has, however, often been considered an epiphenomenon of the underlying pathology. Platelets count alterations are, indeed, usually consensual to other hemogram alterations (anaemia and neutropenia), an indication of a coexisting medullar insufficiency (thrombocytopenia) or other heterogenous diseases such as cancer, iron deficiency or immuno-modulated diseases, usually associated with an increase in comorbidity indexes.12 Those alterations, moreover, can usually influence changes to the therapeutic approach (reduction/suspension of recommended standard therapies) and further condition the prognosis.13 Since a few years, the investigators have been established a cardiac-haematological collaboration aiming at finding early alterations in platelets count or, more generally, in cell blood count (CBC), collegially evaluating those alterations with a cardiologist and a haematologist (even in mild cases) and scheduling, on the basis of the aforementioned evaluations, a more precise and tailored therapeutic approach toward the specific patient needs in order to minimize the downgrading of potentially life-saving therapies.14 Until now, however, no precise evaluation of the impact that this strategy had in influencing the therapeutic approach and in improving patient outcome in our population has been performed.

A retrospective evaluation of consecutive ACS patients, their clinical, biohumoral and procedural characteristics and the adopted pharmacological treatments is, therefore, an important epidemiologic tool for the characterization of this phenomenon and for identifying potential associations which could suggest possible future therapeutic developments.

DETAILED DESCRIPTION:
Even the invasive treatment of coronaropathy during hospitalization, with angioplasty and stent implantation procedures and/or the eventual implantation of temporary mechanical blood circulation assistant devices [aortic counterpulsation, Impella, ECMO (Extracorporeal Membrane Oxygenation)], could further favour the phenomenon. Vice versa, thrombocytosis occurring during ACS has a reactive origin, caused by increased IL-6 production which, in turn, leads to an increase in thrombopoietin formation in the liver, causing a consequent stimulatory activity on megakaryocytes. Different studies have demonstrated a significant correlation between platelets count disorders and patient outcome (survival during hospitalization and in the immediate follow-up). This association has, however, often been considered an epiphenomenon of the underlying pathology. Platelets count alterations are, indeed, usually consensual to other hemogram alterations (anaemia and neutropenia), an indication of a coexisting medullar insufficiency (thrombocytopenia) or other heterogenous diseases such as cancer, iron deficiency or immuno-modulated diseases, usually associated with an increase in comorbidity indexes. Those alterations, moreover, can usually influence changes to the therapeutic approach (reduction/suspension of recommended standard therapies) and further condition the prognosis. Since a few years,the investigators have been established a cardiac-haematological collaboration aiming at finding early alterations in platelets count or, more generally, in cell blood count (CBC), collegially evaluating those alterations with a cardiologist and a haematologist (even in mild cases) and scheduling, on the basis of the aforementioned evaluations, a more precise and tailored therapeutic approach toward the specific patient needs in order to minimize the downgrading of potentially life-saving therapies. Until now, however, no precise evaluation of the impact that this strategy had in influencing the therapeutic approach and in improving patient outcome in our population has been performed.

A retrospective evaluation of consecutive ACS patients, their clinical, biohumoral and procedural characteristics and the adopted pharmacological treatments is, therefore, an important epidemiologic tool for the characterization of this phenomenon and for identifying potential associations which could suggest possible future therapeutic developments.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive ACS subjects hospitalized in the Cardiology 1 - UTIC department of ASST Grande Ospedale Metropolitano Niguarda between 2014 and 2017

Exclusion Criteria:

* Age <18 years
* Subjects admitted with ACS diagnosis but not confirmed at discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Acute Coronary Syndrome diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
net adverse clinical events NACE | 2014 to 2017
  the composite of a list of clinical events

SECONDARY OUTCOMES:
death | 2014 to 2017
  patient's death for all causes at follow up
hospitalization | 2014 to 2017
  duration of patient's hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Opsedaliera Ospedale Niguarda Ca' Granda, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- [Background] Morici N, Tavecchia GA, Antolini L, Caporale MR, Cantoni S, Bertuccio P, Sacco A, Meani P, Viola G, Brunelli D, Oliva F, Lombardi F, Segreto A, Oreglia JA, La Vecchia C, Cattaneo M, Valgimigli M, Savonitto S. Use of PRECISE-DAPT Score and Admission Platelet Count to Predict Mortality Risk in Patients With Acute Coronary Syndrome. Angiology. 2019 Oct;70(9):867-877. doi: 10.1177/0003319719848547. Epub 2019 May 14. PMID 31088127